CLINICAL TRIAL: NCT06612190
Title: Evaluation on Visual Outcome of Transcranial Magnetic Stimulation
Brief Title: Evaluation on Visual Outcome of TMS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Evidence Based Cataract Study Group (Other)
Responsible Party: Principal Investigator, xiangjiazhu, MD, PhD, Evidence Based Cataract Study Group
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EBCSG2024015
Record Dates: First submitted 2024-09-21; First posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Visual Impairment
MeSH Terms: conditions — Vision Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TMS (Experimental)
  Interventions: Procedure: TMS
- Control (Sham Comparator)
  Interventions: Procedure: Control

INTERVENTIONS:
Procedure: TMS — TMS treatment in this study indicates a non-invasive procedure called transcranial magnetic simulation (TMS) on visual cortex. The treatment intensity is set as 80% of the threshold of each participant. The treatment will be conducted every day for consecutive 5 days.
  Arms: TMS
Procedure: Control — The sham group will be given no real magnetic stimulation.
  Arms: Control

SUMMARY:
The goal of this clinical trial is to learn if transcranial magnetic stimulation (TMS) can improve the visual outcomes in patients with visual impairment. The main question it aims to answer is:

• Does TMS improve the visual outcome in patients who suffer from visual impairment? Researchers will compare TMS to the control group who will not receive effective TMS treatment) to see if TMS works to improve the visual outcomes of the patients.

Participants will

* Undergo TMS treatment or no effective TMS for consecutive 5 days.
* Visit the clinic once every 2 weeks for checkups and tests.

ELIGIBILITY:
Inclusion Criteria:

* Post cataract surgery or clear lens
* Best-corrected visual acuity less than 0.1logMAR

Exclusion Criteria:

* Diagnosed with cognitive impairment or mental disorders and unable to cooperate with treatment;
* Diagnosed with ocular diseases that affect observation of visual function;
* History of epileptic seizures;
* Long term use of psychotropic drugs；
* Metal implants in the body.

Ages: 6 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Visual acuity | From enrollment to the end of treatment at 6 months

SECONDARY OUTCOMES:
Visual field | From enrollment to the end of treatment at 6 months

OTHER OUTCOMES:
Visual quality | From enrollment to the end of treatment at 6 months
  Include objective visual quality (contrast sensitivity) and subjective visual quality (visual function questionnaire score).

CONTACTS AND LOCATIONS:
Overall Officials: Xiangjia Zhu, Study Chair — Eye and ENT Hospital of Fudan University; Yating Tang, Principal Investigator — Eye and ENT Hospital of Fudan University; Yinglei Zhang, Principal Investigator — Eye and ENT Hospital of Fudan University; Jiaqi Meng, Principal Investigator — Eye and ENT Hospital of Fudan University; Xin Liu, Principal Investigator — Eye and ENT Hospital of Fudan University
Locations (1):
- Eye and Ear, Nose Throat Hospital of Fudan University, Shanghai, Shanghai Municipality, China